CLINICAL TRIAL: NCT05249907
Title: The Effects of Vibration and Instrument Assisted Soft Tissue Manipulation Methods on Pain and Sleep Quality in Hemodialysis Patients With Restless Legs Syndrome
Brief Title: Hemodialysis Patients With Restless Legs Syndrome Used Vibration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Gülay Turgay, Assist. Prof., Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GTurgay
Record Dates: First submitted 2021-12-09; First posted 2022-02-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-02

CONDITIONS: RLS
Keywords: Hemodialysis; Restless leg sendrome; Vibration; Massage
MeSH Terms: interventions — Massage; Vibration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No application will be made this group
- VIBRATION GROUP (Experimental): Vibration will be applied this group.
  Interventions: Other: Massage
- MASSAGE GROUP (Experimental): Massage will be applied this group.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — Stroking ("stroking") movement will be performed on the soft tissue parallel to the muscle fibers on the origo and insertion lines. Vaseline will be preferred as an intermediate to increase the lubricity of the instrument. The frequency of patting and friction movements will be 60 repetitions per minute.
  Starting from the medial side of the gastrocnemius (calf) muscle in both legs and moving it longitudinally from distal to proximal and from back to distal in a straight line within 20 seconds, for 2.5 minutes. Then this treatment will be applied to the lateral side of the gastrocnemius muscle for 2.5 minutes.
  Other Names: Vibration
  Arms: MASSAGE GROUP; VIBRATION GROUP

SUMMARY:
Restless Legs Syndrome (RLS) is a chronic disorder characterized by abnormal sensations, usually accompanied by pain and restlessness in the legs and/or any part of the body. Sleep quality disorders (10-20%) and limb movements during sleep are quite common in patients with RLS . These disorders in sleep quality are also common among patients receiving hemodialysis due to end-stage renal disease.

Pharmacological and non-pharmacological methods are used in the treatment of RLS.

Due to the varying success and side effects of pharmacological treatments, non-pharmacological methods have come to the fore for these patients. One of the methods that can be applied as a non-pharmacological method is vibration.

The therapeutic effect of instrument-assisted soft tissue manipulation (EYYDM) is not clear, it is stated that it activates the muscles, fascia and tendon and improves pain clinically in studies.

The aim of the study is to determine the most effective treatment method on pain and sleep quality by comparing the effects of vibration and EYYDM methods in dialysis patients with restless legs syndrome

DETAILED DESCRIPTION:
Restless Legs Syndrome (RLS) is a chronic disorder characterized by abnormal sensations, usually accompanied by pain and restlessness in the legs and/or any part of the body. The typical clinical feature of RLS is the irresistible urge to move and restlessness, especially in the legs, that prevents falling asleep, accompanied by dysesthesia, and the symptoms are more pronounced in the evening and at night, and occur and increase at rest.

Sleep quality disorders (10-20%) and limb movements during sleep are quite common in patients with RLS . These disorders in sleep quality are also common among patients receiving hemodialysis due to end-stage renal disease.

Pharmacological and non-pharmacological methods are used in the treatment of RLS.

Due to the varying success and side effects of pharmacological treatments, non-pharmacological methods have come to the fore for these patients. One of the methods that can be applied as a non-pharmacological method is vibration. Vibration causes an increase in the patient's body temperature, leading, in turn, to increased oxygen release from myoglobin and hemoglobin, increased muscle blood flow, increased sensitivity of neural receptors, increased nerve velocity, and decreased muscle viscosity. It has been stated that all these factors contribute positively to improving health, reducing pain, improving sleep quality, as well as bio-motor and functional indicators.

Although the therapeutic effect of instrument-assisted soft tissue manipulation (EYYDM) is not clear, it is stated that it activates the muscles, fascia and tendon and improves pain clinically in studies.

In Turkey, no study investigating the effects of vibration and EYYDM in hemodialysis patients diagnosed with RLS has been found. In this direction, the aim of the study is to determine the most effective treatment method on pain and sleep quality by comparing the effects of vibration and EYYDM methods in dialysis patients with restless legs syndrome

ELIGIBILITY:
Inclusion Criteria:

Receiving hemodialysis treatment for at least 6 months 3 days a week for 4 hours Patients with RLS according to the diagnostic criteria of the International RLS study group In laboratory examinations the kinetic indicators of dialysis adequacy are within the desired target range (Kt/V: 1.2-1.3; URR: 60-65%) radiological examinations without pathological findings (fracture, dislocation, tumor, infection)

Exclusion Criteria:

psychiatric problems neurological deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Massage Group | 1 month
  Massage will applied for three day a week
Vibration Group | 1 month
  Vibration will applied for three day a week
Sleep quality | 1 month later
  Sleep quality of the patients will be measured with the pittsburg sleep quality scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Gülşen, Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Article
Supporting Information: CSR
Time Frame: with in a year
Access Criteria: pubmed